CLINICAL TRIAL: NCT07201168
Title: Impact of a Structured Multimodal Educational Program on Clinical Outcomes and Quality of Life in Patients With Critical Limb Ischemia: A Randomized Controlled Trial.
Brief Title: Structured Educational Program vs Standard Care in Pre-surgical Critical Limb Ischemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulip Medicine (Other)
Responsible Party: Principal Investigator, Didar Khassenov, Head of department, Tulip Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NROC 3
Record Dates: First submitted 2025-09-17; First posted 2025-10-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Health Education
Keywords: critical limb ischemia; peripheral artery disease; patient education; structured education program; quality of life; chronic limb threatening ischemia; health education; randomized controlled trial
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Program + Standard Medical Care (Experimental): Participants receive a comprehensive 4-week multimodal educational program including interactive group sessions, digital platform access, printed materials, and medical hotline access in addition to standard medical care.
  Interventions: Other: Structured Multimodal Educational Program for Critical Limb Ischemia
- Standard Medical Care (Other): Participants receive standard medical care for critical limb ischemia including routine vascular surgery consultation, standard medical management, and usual wound care instructions without any structured educational intervention.
  Interventions: Other: Standard medical care

INTERVENTIONS:
Other: Structured Multimodal Educational Program for Critical Limb Ischemia — A comprehensive 4 weeks educational program combining face-to-face and digital learning modalities. Components include: interactive group sessions twice a week led by vascular specialists covering the pathophysiology of disease, risk factor modification, and treatment options; digital platform access with multimedia educational materials, printed educational materials for home reference; peer support group participation; medical hotline access for patient-initiated consultations and urgent questions; smoking cessation counseling; supervised exercise program recommendations; wound care training. The program emphasizes patient self-management skills, early recognition of complications, and adherence to medical therapy alongside standard clinical care.
  Arms: Educational Program + Standard Medical Care
Other: Standard medical care — Routine clinical management for critical limb ischemia according to current standard of care guidelines. Includes vascular surgery consultation and scheduled follow-up appointments as clinically indicated. No structured educational materials, formal patient education sessions, or additional follow-up contacts beyond routine clinical care are provided. Patients receive standard verbal and written instructions during consultation and have access to the same medical and surgical treatments as the intervention group when clinically warranted.
  Arms: Standard Medical Care

SUMMARY:
Critical limb ischemia (CLI) is a severe condition where poor blood flow to the legs causes pain, non-healing wounds, and may require amputation. It affects 10% of people over 40, rising to 20% in those over 70. Within the first year after diagnosis, 30% of patients need amputation and 25% die.

Current treatments include medications, surgery to restore blood flow, or amputation, but results remain poor. Research shows that lifestyle changes like quitting smoking and regular exercise can significantly improve outcomes, yet most CLI patients struggle to make these changes and lack knowledge about their condition.

This study tests whether a structured educational program called the "Critical Limb Ischemia School" can help patients. The program teaches patients about their condition, symptom management, lifestyle modifications, and when to seek medical help. The investigators will compare patients receiving this education to those getting standard care.

The study will evaluate several important health outcomes during a 12-month period to determine if the educational program makes a meaningful difference in patients' lives. The investigators will assess how the intervention affects patients' overall well-being, their ability to manage symptoms and daily activities, and whether it helps prevent serious complications that could lead to disability.

If successful, this program could provide a cost-effective way to help CLI patients manage their condition and potentially avoid serious complications like amputation.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the effectiveness of a structured multimodal educational program (School of Critical Limb Ischemia) compared to standard medical care in improving clinical outcomes for patients with critical limb ischemia (CLI).

Modifiable risk factors including smoking, physical inactivity, uncontrolled diabetes, hypertension, and dyslipidemia play crucial roles in disease progression. Research demonstrates that comprehensive risk factor modification significantly improves outcomes-patients who quit smoking have 14% five-year mortality compared to 31% among continued smokers. Despite this evidence, patient adherence remains low, with only 5-30% successfully quitting smoking and fewer than 50% engaging in recommended exercise programs.

Educational interventions have proven effective in other chronic conditions such as diabetes and heart failure, improving patient self-management and clinical outcomes. However, significant knowledge gaps exist among CLI patients-only 54% are aware of multiple treatment options, 24% incorrectly believe no additional treatment is needed after surgery, and only 31% understand the priority of conservative therapy over invasive interventions. This highlights the critical need for structured educational programs specifically designed for CLI patients.

The intervention combines traditional face-to-face education with digital technologies to create a personalized, accessible learning experience addressing disease understanding, risk factor modification, symptom recognition and management, and shared decision-making. The program utilizes interactive group sessions, individual counseling, digital platforms with multimedia materials, printed resources, peer support, and regular follow-up contact. Participants are randomly assigned to receive either the educational program plus standard medical care or standard medical care alone, with 12-month follow-up to assess both short-term and medium-term outcomes.

If successful, this research could transform CLI management by providing evidence for implementing structured educational programs in vascular surgery practices. Given the substantial economic burden of CLI treatment (estimated at USD 24,000-72,000 per patient in the first year), even modest improvements in clinical and economic outcomes could result in significant healthcare cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of chronic critical limb ischemia (CLI)
* Rutherford category 2-5
* Ability to understand study procedures and provide signed and dated written informed consent
* Fluency in Russian language
* Access to telephone and internet

Exclusion Criteria:

* Severe cognitive impairment
* Participation in another clinical trial that might interfere with study outcomes
* Planned major amputation within 3 months
* Diabet 1 and 2 type
* Inability to attend scheduled educational sessions
* Severe visual or hearing impairments that would interfere with participation in educational sessions
* Patients who declined to participate after being informed about the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Frequency of CLI-related hospitalizations | 12 months from enrollment
  Total number of hospitalizations related to critical limb ischemia or its complications (such as limb infections, need for revascularization, amputation) per patient during the follow-up period.
SF-12 Quality of Life Score | Baseline, 6 months, and 12 months from enrollment
  12-Item Short Form Health Survey (SF-12) Physical Component Summary (PCS): 0-100 Mental Component Summary (MCS): 0-100 Higher scores indicate better quality of life and better health status.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Baseline, 6 months, and 12 months from enrollment
  Pain intensity assessed using the Visual Analog Scale (VAS). Score range: 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores indicate worse pain.
Proportion of disability cases | 12 months from enrollment
  Percentage of new disability cases or changes in disability status during the follow-up period.
Smoking cessation rate | 12 months from enrollment
  Percentage of patients who successfully quit smoking at 12 months follow-up among those who were smokers at baseline, defined as self-reported abstinence from smoking in the past month.
Pain-free walking distance | Baseline, 12 months from enrollment
  Distance walked before onset of leg pain assessed by smartphone pedometer during standardized walking test at self-selected comfortable pace until onset of claudication pain.
Quality-Adjusted Life Years (QALY) | 12 months from enrollment
  Health utility measured using SF-6D utility scores derived from SF-12 questionnaire, calculated using the area under the curve method over the 12-month study period The QALY score will range from 0 to 1. A higher QALY score represents a better overall health outcome over the 12-month period, indicating more time spent in a better state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- NCJSC "Astana Medical University", Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No